CLINICAL TRIAL: NCT06142266
Title: Assessment of Improvement in Functional Status in Moderate to Severe Stable COPD Patients After Exercise Rehabilitation Program
Brief Title: Functional Status in COPD Patients After Exercise Rehabilitation Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, Lecture of chest diseases, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COPD&Exercise rehabilitation
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: randomized controlled trial conducted at Chest Department at Assiut University Hospital
Who Masked: Participant
Masking Description: Participants will be randomly allocated to either the intervention or control group in a 1:1 ratio using computer-generated randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group (n=60) will undergo a 12-week pulmonary rehabilitation program. This program will consist of twice-weekly supervised exercise sessions, including aerobic training and resistance exercises targeting the lower limbs.
  Interventions: Other: Exercise rehabilitation program
- Control group (Active Comparator): The control group (n=60) will receive usual medical care according to guidelines, which may include bronchodilator/anti-inflammatory therapy but no formal pulmonary rehabilitation.
  Interventions: Other: Exercise rehabilitation program

INTERVENTIONS:
Other: Exercise rehabilitation program — This program will consist of twice-weekly supervised exercise sessions, including aerobic training and resistance exercises targeting the lower limbs for 12-week

SUMMARY:
To evaluate the effectiveness of the exercise program in improving physical fitness and exercise capacity in COPD patients like walking distance, muscle strength, endurance will be measured before and after the program.

To assess whether the program helps reduce COPD symptoms like shortness of breath and fatigue during daily activities. Quality of life questionnaires will be used.

DETAILED DESCRIPTION:
Pulmonary rehabilitation is a comprehensive, multidisciplinary program that utilizes exercise training and patient education to improve the physical and psychological condition of people living with chronic respiratory diseases Exercise therapy and education work in an integrated manner to help patients better manage their condition.

Exercise therapy is a core component of pulmonary rehabilitation. Regular physical activity helps build endurance, strengthen respiratory muscles, and improve overall functional capacity . Both aerobic and resistance exercises are prescribed according to individual abilities and needs .Studies have shown exercise training can reduce symptoms, increase quality of life, and decrease healthcare utilization among pulmonary patients .Patient education teaches self-management skills like breathing techniques, medication management, coping strategies, and how to prevent or deal with exacerbations . Educating patients empowers them to better understand their condition and play an active role in their care. It also helps address anxiety and depression that often accompany chronic lung disease .

Recent reviews continue to support the benefits of pulmonary rehabilitation's holistic, exercise-education approach meta-analysis found multidisciplinary programs significantly improved outcomes such as hospital admissions compared to usual care . Additionally, study showed telerehabilitation with remote exercise monitoring and video classes achieved comparable benefits to traditional center-based programs . In summary, exercise therapy and education are core components of effective pulmonary rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate-severe chronic obstructive pulmonary disease (COPD) based on spirometry results and clinical assessment.
* Age between 40 and 75 years. Stable disease status, defined as no exacerbations requiring admission to respiratory intensive care unit
* Willingness and ability to participate in a 12-week pulmonary rehabilitation program.

Exclusion Criteria:

* Presence of significant comorbidities or medical conditions that may interfere with participation in the pulmonary rehabilitation program (e.g., severe cardiovascular disease, musculoskeletal disorders, uncontrolled hypertension).
* Inability to perform the required exercise activities due to physical limitations or disabilities.

Cognitive impairment

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in exercise capacity | baseline
  Asess by Change in 6-minute walk distant

SECONDARY OUTCOMES:
Health related quilt of life | baseline
  Asess by St .George Questioner

CONTACTS AND LOCATIONS:
Overall Officials: Heba fahmy, MD, Study Chair — Assiut University

REFERENCES:
- [Background] Gloeckl R, Schneeberger T, Jarosch I, Kenn K. Pulmonary Rehabilitation and Exercise Training in Chronic Obstructive Pulmonary Disease. Dtsch Arztebl Int. 2018 Feb 23;115(8):117-123. doi: 10.3238/arztebl.2018.0117. PMID 29526182
- [Background] Rutkowski S, Rutkowska A, Kiper P, Jastrzebski D, Racheniuk H, Turolla A, Szczegielniak J, Casaburi R. Virtual Reality Rehabilitation in Patients with Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2020 Jan 13;15:117-124. doi: 10.2147/COPD.S223592. eCollection 2020. PMID 32021150